CLINICAL TRIAL: NCT00796822
Title: A Randomized, Placebo-Controlled Trial of Pentoxifylline to Improve Endothelial Function in HIV-Infected Patients Not Requiring Antiretroviral Therapy
Brief Title: Evaluating the Effectiveness of Pentoxifylline at Improving Blood Vessel Function in HIV-infected People Not Receiving Antiretroviral Medications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Samir K Gupta, MD, MS, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 614; R01HL095149 (NIH)
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Results first posted 2013-05-17 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: HIV; Cardiovascular Diseases; Atherosclerosis
Keywords: Endothelial Function; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Inflammation | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive pentoxifylline.
  Interventions: Drug: Pentoxifylline
- 2 (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — 400 mg three times a day for 8 weeks
  Arms: 1
Drug: Placebo — One pill three times a day for 8 weeks
  Arms: 2

SUMMARY:
People infected with HIV have a greater risk of developing cardiovascular disease than people not infected with HIV. This may be due to increased inflammation brought on by either the HIV infection itself or the use of antiretroviral medications to treat HIV infection. This study will evaluate an anti-inflammatory drug, pentoxifylline, to determine whether it improves blood vessel function and reduces inflammation in people infected with HIV who are not currently receiving antiretroviral medications.

DETAILED DESCRIPTION:
People infected with HIV have an increased risk for cardiovascular disease, which is a leading cause of death for those with HIV. The increase in cardiovascular disease has been thought to be linked to the use of several types of antiretroviral medications used to treat HIV infection. These medications have been shown to cause insulin resistance and dyslipidemia, or high cholesterol levels-conditions that can lead to atherosclerosis, which is a build-up of plaque within the arteries, and ultimately to cardiovascular disease. However, new research is emerging that suggests that people infected with HIV who do not receive antiretroviral medications may also have an increased risk of cardiovascular disease as a result of increased endothelial dysfunction. This condition, which involves malfunctioning of the thin layer of cells that line the interior surface of blood vessels, can lead to atherosclerosis and cardiovascular disease. Pentoxifylline is a medication that is currently used to reduce leg pain in people with blockages in the blood vessels in their legs. Previous research has shown that pentoxifylline may reduce inflammation and improve blood vessel function in people infected with HIV, but more research is needed to confirm these benefits. The purpose of this study is to determine whether pentoxifylline reduces inflammation and improves endothelial function in HIV-infected people who are not receiving antiretroviral medications.

This study will enroll HIV-infected people who are not currently receiving antiretroviral medications. At a baseline study visit, participants will undergo a medical history review; physical examination; measurements in blood pressure, heart rate, height, weight, waist, and hip; and blood and urine collection. An ultrasound imaging test of the arm will measure blood vessel function. Participants will then be randomly assigned to receive either pentoxifylline or placebo three times a day for 8 weeks. At study visits at Weeks 4 and 8, participants will undergo repeat baseline measurements.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of HIV infection with a positive HIV enzyme-linked immunosorbent assay (ELISA) test and confirmatory western blot test
* CD4 cell count greater than 350/µL at the time of screening
* Has not received any antiretroviral therapies in the 6 months before screening
* No anticipated need for any antiretroviral therapies during the course of this study, as determined by the principal investigator or by the participant's HIV caregiver

Note: There is no HIV-1 RNA level eligibility criterion.

Exclusion Criteria:

* Incarceration at the time of screening or at any study visit
* Diagnosed vascular disease, including history of angina pectoris, coronary disease, peripheral vascular disease, cerebrovascular disease, aortic aneurysm, or otherwise known atherosclerotic disease
* Diagnosed disease or process, other than HIV infection, associated with increased systemic inflammation (including, but not limited to, systemic lupus erythematosis, inflammatory bowel diseases, or other collagen vascular diseases). Hepatitis B or C co-infections are NOT exclusionary.
* History of bleeding diathesis, gastrointestinal ulceration or bleeding, cerebrovascular aneurysm or bleeding, or retinal hemorrhage
* Known or suspected cancer requiring systemic treatment in the 6 months before screening
* History of American Diabetes Association (ADA)-defined diabetes mellitus. History of gestational diabetes is not exclusionary if the potential participant does not have current ADA-defined diabetes.
* History of migraine headaches
* History of Raynaud's phenomenon
* History of cardiac arrhythmias or cardiomyopathy
* History of hypothyroidism or hyperthyroidism, even if treated
* Known allergy or intolerance to pentoxifylline or other methylxanthines (e.g., theophylline, caffeine, theobromine). Use of caffeinated products, except on the mornings of the study visits, is not exclusionary.
* Known allergy or intolerance to nitroglycerin
* History of carotid bruits
* Creatinine clearance less than 50 mL/min, using the Cockcroft-Gault equation and a serum creatinine level measured in the 28 days before screening or at the screening visit
* Hemoglobin less than 9.0 mg/dL in the 28 days before screening or at the screening visit
* Alanine aminotransferase (ALT) level or aspartate aminotransferase (AST) greater than three times the upper limit of normal (ULN) in the 28 days before screening or at the screening visit
* Total bilirubin greater than 2.5 times the ULN in the 28 days before screening or at the screening visit
* Fever, defined as a temperature greater than or equal to 38.0 C in the 48 hours before screening. Fever in the 48 hours before each study visit will require postponement of that study visit until the participant's temperature has been lower than 38.0 C for at least 48 hours; fevers continuing past the allowed study visit timeframe will result in study discontinuation.
* Therapy for acute infection or other serious medical illnesses in the 14 days before screening. Therapy for acute infection or other serious medical illnesses that overlaps with a study visit will result in postponement of that study visit until the course of therapy is completed; postponement outside of the allowed study visit timeframe will result in study discontinuation.
* Pregnant or breastfeeding
* Hypotension, defined as systolic blood pressure less than 90 mm Hg, at time of screening. Hypotension noted prior to brachial artery reactivity testing at each study visit will result in study visit postponement of at least 1 day until systolic pressure is greater than or equal to 90 mm Hg the morning of brachial reactivity testing; postponement outside of the allowed study visit timeframe will result in study discontinuation.
* Hypertension, defined as the receipt of any antihypertensive medication in the 28 days before screening or systolic blood pressure greater than 160 mm Hg at the screening visit
* Receipt of anti-inflammatory agents (including, but not limited to, plaquenil, infliximab, etanercept, mycophenolate mofetil, sirolimus, tacrolimus, cyclosporine, pentoxifylline, or thalidomide) in the 28 days before screening
* Receipt of investigational agents, cytotoxic chemotherapy, systemic or topical glucocorticoids (of any dose), or anabolic steroids in the 28 days before screening. Physiologic testosterone replacement therapy is not exclusionary.
* Receipt of lipid-lowering drugs, aspirin, other non-steroidal anti-inflammatory drugs (NSAIDS), acetazolamide, anticoagulants, anticonvulsants, or thyroid replacements in the 28 days before screening
* Use of sildenafil, vardenafil, or tadalafil in the 72 hours before or after each study visit
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir K. Gupta, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana Clinical Research Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Gupta SK, Mi D, Dube MP, Saha CK, Johnson RM, Stein JH, Clauss MA, Mather KJ, Desta Z, Liu Z. Pentoxifylline, inflammation, and endothelial function in HIV-infected persons: a randomized, placebo-controlled trial. PLoS One. 2013 Apr 9;8(4):e60852. doi: 10.1371/journal.pone.0060852. Print 2013. PMID 23593327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment, enrollment, and follow-up assessments were performed from May 2009 through October 2011, at the HIV outpatient clinics of the Indiana University Health medical system.
Pre-assignment Details: Potential participants underwent a screening visit to evaluate eligibility within 21 days of randomization.
Groups:
- Pentoxifylline: Participants will receive pentoxifylline.
  Pentoxifylline : 400 mg three times a day for 8 weeks
- Placebo: Participants will receive placebo.
  Placebo : One pill three times a day for 8 weeks
Period: Overall Study
Arm/Group | Pentoxifylline | Placebo
Started | 13 | 13
Completed | 10 | 13
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10.9) | 40 (11.6) | 37 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow-mediated Dilation of the Brachial Artery
Description: Flow-mediated dilation is nn in vivo measure of arterial endothelial function. We assessed changes in flow-mediated dilation from baseline to week 8.
Time Frame: Measured at baseline and Week 8
Population: Number of remaining participants at week 8 with evaluable vascular ultrasonography. In the Pentoxifylline group, 10 participants were evaluated at week 8 but only 9 had evaluable ultrasonography.
Measure: Mean (Standard Deviation); unit: absolute percentage
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 9 | 13
absolute percentage | -1.93 (3.03) | -1.06 (1.45)
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; The sample size was determined based on a two-sample, independent, two-tailed t-test with 5% type I error. Using the results from our pilot trial, we conservatively estimated a predicted absolute change in FMD of 3.5% with PTX (assuming no change with placebo) and we assumed a common standard deviation of 2.6%. A sample size of 10 per group was estimated to provide at least 80% power to detect this effect size. Allowing for a 20% dropout rate, we planned to recruit 13 subjects per group; Test type: Superiority or Other; p = 0.44, t-test, 2 sided; Mean Difference (Net) = -0.87, 95% CI 2-sided [-1.53 to 3.28], Standard Deviation 1.09

2. Secondary Outcome: Change in Soluble TNF-Receptor I Levels
Description: Measure of systemic inflammation
Time Frame: Measured at baseline and Week 8
Population: Those who had both baseline and Week 8 data available
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 10 | 13
pg/mL | 65.9 (168.97) | -83.2 (137.45)
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Test type: Superiority — There was no formal power calculation for this outcome measure as the study was powered on the primary outcome measure; p = 0.03, t-test, 2 sided; Median Difference (Net) = 149.1, 95% CI 2-sided [16.4 to 281.9], Standard Deviation 151.8

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Pentoxifylline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 10/13 | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentoxifylline (N=13) | Placebo (N=13)
All gastrointestinal (Gastrointestinal disorders) | 5 (7) | 5 (8) — Nausea, vomiting, belching, dyspepsia, diarrhea
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Headache (General disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypokalemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyperkalemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Elevated liver function tests (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No